CLINICAL TRIAL: NCT02001701
Title: Intravitreal Injection of Expansile Sulfa Hexafluoride Gas for Symptomatic Vitreomacular Adhesion
Brief Title: Intravitreal Gas for Vitreomacular Adhesion
Acronym: RELEASE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were enrolled.
Sponsor: Northern California Retina Vitreous Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCRVA - 2013 - RELEASE
Record Dates: First submitted 2013-11-24; First posted 2013-12-05 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Vitreomacular Adhesion
Keywords: vitreomacular adhesion; vitreomacular traction; macular hole; epiretinal membrane; intravitreal gas; sulfahexafluoride gas; perfluoropropane gas; ocriplasmin; vitrectomy
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Gas (Experimental): Intravitreal injection of sulfahexafluoride gas
  Interventions: Procedure: Intravitreal Injection of sulfahexafluoride gas

INTERVENTIONS:
Procedure: Intravitreal Injection of sulfahexafluoride gas — After the appropriate sterile and anesthetic preparation of the surgical field, the investigator will administer a single intravitreal injection of 0.3 to 0.5 cc of sulfahexafluoride gas in the study eye. An anterior chamber paracentesis may be performed if necessary. Following the procedure, the optic nerve will be monitored for perfusion.

SUMMARY:
Vitreomacular adhesion causes symptoms of blurry vision, distortion, and double vision. It is due to an abnormal separation of the vitreous gel from the surface of the retina and macula. The current, gold-standard treatment for this condition involves surgery performed in the operating room that involves risk such as bleeding, infection, cataract, and retinal detachment. It has been previously shown that a less invasive intravitreal injection of a gas bubble performed in the office may also treat vitreomacular adhesion with less risk than surgery.

The purpose of this study is to determine the effect of an office-based injection of an intravitreal gas bubble as a treatment for symptomatic vitreomacular adhesion.

DETAILED DESCRIPTION:
Symptomatic vitreomacular adhesion (sVMA), also known as Vitreomacular traction (VMT) is thought to occur due to an anomalous or incomplete posterior vitreous detachment (PVD).1 Typical symptoms of VMT include decreased reading vision and metamorphopsia. Ultra-high resolution spectral-domain optical coherence tomography (SD-OCT) has greatly enhanced our understanding of the spectrum of the vitreomacular interface disorders ranging from focal adhesions, macular cysts, impending macular holes, full thickness macular holes, lamellar holes, and epiretinal membrane.2 Generally, pars plana vitrectomy (PPV) surgery is the preferred treatment for many of these conditions with high success rates.3 However, surgical intervention is not without risk and includes the potential for infection, retinal detachment, cataract progression, and patient discomfort from post-operative prone positioning in cases of macular hole.4 Despite the high success rate with vitrectomy, the risks of surgery have led researchers to search for non-surgical treatments of VMT such as pharmacologic vitreolysis. Ocriplasmin (JetreaTM, ThromboGenics, Inc. Iselin, NJ) was recently approved by the United States Food & Drug Administration (FDA) in October 2012 as a non-surgical, pharmacologic agent for the treatment of symptomatic VMA.5 Pooled data from two phase III clinical trials of ocriplasmin (MIVI-TRUST)5 demonstrated that approximately 26% of eyes treated with a single intravitreal injection of ocriplasmin (125 ug) compared to 10% of eyes treated with vehicle alone (placebo) resulted in resolution of VMA on OCT at 28 days. Potential side effects of ocriplasmin include transient floaters, zonular instability, and transient vision loss.6 Although the primary outcome of the study achieved a statistically significant result compared to placebo, the less than robust results compared to surgical intervention with the associated high cost of the medication have led retina specialists to question the clinical utility of this medication.

Previous small case series' have demonstrated that an intravitreal gas bubble injection alone (i.e. pneumatic vitreolysis) may lead to macular hole closure through the induction of a PVD.7-9 Additional small cases series' have shown that an intravitreal gas bubble alone may induce a PVD in patients with non-proliferative diabetic retinopathy10 and diabetic macular edema11 in nearly 100% of cases. One small case series showed that an intravitreal gas bubble in combination with an anti-vascular endothelial growth factor agent can cause resolution of VMA in patients with wet macular degeneration in 4/4 (100%) of eyes.12 However, there is a paucity of literature on the specific treatment of isolated VMT with intravitreal gas alone. Recently, Rodriques et al13 demonstrated that a single intravitreal injection of perfluoropropane (C3F8) gas injection may cause VMT resolution in 5/7 (70%) eyes with isolated VMT and in 3/6 (50%) eyes with diabetic macular edema. Although this initial study demonstrated efficacy, the overall success rate of the procedure as well as the visual acuity benefit was limited due to the heterogeneous patient population. Pneumatic vitreolysis may offer a potential safe, low cost, and effective procedure that may pose an alternative to treatment in patients with symptomatic vitreomacular adhesion.

The purpose of the present study is to evaluate the efficacy and safety of the administration of a single intravitreal injection of sulfa hexafluoride (SF6) gas for patients with symptomatic vitreomacular adhesion without concomitant macular hole. Key differences between the present study and that by Rodriques et al.10 are the use of a shorter acting gas bubble (SF6 vs C3F8) and the inclusion of a homogenous patient population with VMA alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide written informed consent
* Patients with Symptomatic Vitreomacular Adhesion (sVMA) as defined by Clinical and SD-OCT findings:
* Clinical Findings:

  1. Symptoms: blurred vision, double vision, metamorphopsia, micropsia
  2. Snellen Visual Acuity: < 20/25 in study eye
* SD-OCT (Cirrus, Car Zeiss Meditec, Dublin, CA) Findings:

  1. Visible vitreous attachment within a 1,500 um radius of the foveal center causing antero-posterior vitreofoveal traction with associated microstructural retinal changes
  2. See Figure 1 (Image "E") for representative candidates for inclusion.
* Observation period of 1 month prior to intervention allowing for spontaneous resolution

Exclusion Criteria:

* Figure 1 (Images "A", "B", "C", "D", "F", "H", "I")
* Any Macular Hole
* Epiretinal Membrane
* History of Diabetic Retinopathy (non-proliferative, proliferative, and/or diabetic macular edema)
* Macular Degeneration
* Retinal vascular occlusion
* Aphakia
* High myopia (> -8 diopters)
* Uncontrolled glaucoma
* Vitreous Opacification
* Retinal tear or retinal detachment
* Vitrectomy surgery
* Macular laser

Figure 1: Refer to the following article:

Stalmans P, Duker JS, Kaiser PK, et al. OCT-Based Interpretation of the Vitreomacular Interface and Indications for Pharmacologic Vitreolysis. Retina; 2013: Epub ahead of print

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with resolution of vitreomacular adhesion at Day 28 | Day 28

SECONDARY OUTCOMES:
Change in Visual Acuity | Day 14
Change in Visual Acuity | Day 28
Change in Visual Acuity | Day 90
Time to resolution of vitreomacular adhesion | Day 90
Proportion of patients requiring vitrectomy surgery | Day 90
  The investigator may consider vitrectomy surgery if:
  1. Decrease in Visual Acuity
  2. Worsening of vitreomacular adhesion on SD-OCT
  3. Progression of vitreomacular adhesion to macular hole
  4. No improvement of vitreomacular adhesion by Day 28
Incidence of Retinal Tears and Retinal Detachment | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Alok S Bansal, MD, Principal Investigator — Northern California Retina Vitreous Associates
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stalmans P, Duker JS, Kaiser PK, Heier JS, Dugel PU, Gandorfer A, Sebag J, Haller JA. Oct-based interpretation of the vitreomacular interface and indications for pharmacologic vitreolysis. Retina. 2013 Nov-Dec;33(10):2003-11. doi: 10.1097/IAE.0b013e3182993ef8. PMID 23881226
- [Background] Chang LK, Fine HF, Spaide RF, Koizumi H, Grossniklaus HE. Ultrastructural correlation of spectral-domain optical coherence tomographic findings in vitreomacular traction syndrome. Am J Ophthalmol. 2008 Jul;146(1):121-7. doi: 10.1016/j.ajo.2008.03.001. Epub 2008 Apr 25. PMID 18439563
- [Background] Witkin AJ, Patron ME, Castro LC, Reichel E, Rogers AH, Baumal CR, Duker JS. Anatomic and visual outcomes of vitrectomy for vitreomacular traction syndrome. Ophthalmic Surg Lasers Imaging. 2010 Jul-Aug;41(4):425-31. doi: 10.3928/15428877-20100525-07. Epub 2010 May 28. PMID 20608611
- [Background] Recchia FM, Scott IU, Brown GC, Brown MM, Ho AC, Ip MS. Small-gauge pars plana vitrectomy: a report by the American Academy of Ophthalmology. Ophthalmology. 2010 Sep;117(9):1851-7. doi: 10.1016/j.ophtha.2010.06.014. PMID 20816248
- [Background] Stalmans P, Benz MS, Gandorfer A, Kampik A, Girach A, Pakola S, Haller JA; MIVI-TRUST Study Group. Enzymatic vitreolysis with ocriplasmin for vitreomacular traction and macular holes. N Engl J Med. 2012 Aug 16;367(7):606-15. doi: 10.1056/NEJMoa1110823. PMID 22894573
- [Background] Freund KB, Shah SA, Shah VP. Correlation of transient vision loss with outer retinal disruption following intravitreal ocriplasmin. Eye (Lond). 2013 Jun;27(6):773-4. doi: 10.1038/eye.2013.94. Epub 2013 May 3. No abstract available. PMID 23640609
- [Background] Chan CK, Wessels IF, Friedrichsen EJ. Treatment of idiopathic macular holes by induced posterior vitreous detachment. Ophthalmology. 1995 May;102(5):757-67. doi: 10.1016/s0161-6420(95)30958-x. PMID 7777275
- [Background] Jorge R, Costa RA, Cardillo JA, Uno F, Bonomo PP, Farah ME. Optical coherence tomography evaluation of idiopathic macular hole treatment by gas-assisted posterior vitreous detachment. Am J Ophthalmol. 2006 Nov;142(5):869-71. doi: 10.1016/j.ajo.2006.05.062. PMID 17056375
- [Background] Mori K, Saito S, Gehlbach PL, Yoneya S. Treatment of stage 2 macular hole by intravitreous injection of expansile gas and induction of posterior vitreous detachment. Ophthalmology. 2007 Jan;114(1):127-33. doi: 10.1016/j.ophtha.2006.07.001. Epub 2006 Oct 27. PMID 17070585
- [Background] Ochoa-Contreras D, Delsol-Coronado L, Buitrago ME, Velasco-Barona C, Quiroz-Mercado H. Induced posterior vitreous detachment by intravitreal sulfur hexafluoride (SF6) injection in patients with nonproliferative diabetic retinopathy. Acta Ophthalmol Scand. 2000 Dec;78(6):687-8. doi: 10.1034/j.1600-0420.2000.078006687.x. PMID 11167234
- [Background] McHugh D, Gupta B, Saeed M. Intravitreal gas injection for the treatment of diabetic macular edema. Clin Ophthalmol. 2011;5:1543-8. doi: 10.2147/OPTH.S25348. Epub 2011 Oct 26. PMID 22125399
- [Background] Kim YM, Lee SJ, Koh HJ. Gas-assisted release of vitreomacular adhesion in wet age-related macular degeneration. Retina. 2011 Nov;31(10):2123-4. doi: 10.1097/IAE.0B013E31822F5720. No abstract available. PMID 22027799
- [Background] Rodrigues IA, Stangos AN, McHugh DA, Jackson TL. Intravitreal injection of expansile perfluoropropane (c(3)f(8)) for the treatment of vitreomacular traction. Am J Ophthalmol. 2013 Feb;155(2):270-276.e2. doi: 10.1016/j.ajo.2012.08.018. Epub 2012 Nov 17. PMID 23164159
- See also: Northern California Retina Vitreous Associates — http://www.ncrva.com